CLINICAL TRIAL: NCT03259204
Title: Prevention of Thromboembolism and Failed Healing During Lower Limb Immobilization - Multicenter Study With Adjuvant Intermittent Pneumatic Compression Therapy
Brief Title: Swedish Multicenter Trial of Outpatient Prevention of Leg Clots
Acronym: StopLegClots
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Sahlgrenska University Hospital (Other); Danderyd Hospital (Other); Stockholm South General Hospital (Other); Uppsala University Hospital (Other); Gävle Hospital (Other); Höglandssjukhuset Eksjö (Unknown); Norrtälje Hospital (Unknown); Östersund Hospital (Unknown); Helsingborgs Hospital (Other); Uddevalla Hospital (Unknown); Norra Älvsborgs Länssjukhus (Unknown); Istituto Ortopedico Rizzoli (Other); Lugano Regional Hospital (Unknown); Alingsås Lasarett (Unknown); University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Paul Ackermann, Professor, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017-00202
Record Dates: First submitted 2017-08-16; First posted 2017-08-23 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Achilles Tendon Rupture; Ankle Fractures; Venous Thromboembolism
Keywords: Achilles tendon; Microdialysis; Immobilization; Wound healing; Intermittent Pneumatic Compression; Ultrasonography
MeSH Terms: conditions — Ankle Fractures; Venous Thromboembolism

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leg Immobilization (No Intervention): Routine care include that the lower limb will be immobilized in an orthosis or a below-knee plaster cast according to local routines.
- Adjuvant IPC (Experimental): Leg Immobilization with the addition of IPC. Patients will during lower limb immobilization receive bilateral calf IPC.
  Interventions: Device: Adjuvant IPC

INTERVENTIONS:
Device: Adjuvant IPC — This IPC-system delivers sequential circumferential compression. The IPC device is mobile and should therefore not restrict patient mobilization, but can be taken off if the patient wants to mobilize independently.
  Arms: Adjuvant IPC

SUMMARY:
Lower limb immobilization is associated with high risk of complications, i.e. venous thromboembolism (VTE) and failed healing. Pharmacoprophylaxis of VTE is in leg-immobilized patients, however, low- or non-effective and associated with adverse events. Thus, there is a need for novel treatments.

This study aims to demonstrate in leg immobilized patients who have suffered an ankle fracture (1000 patients) or an Achilles tendon rupture (400 patients) that adjuvant intermittent pneumatic compression (IPC) therapy, which targets impaired vascular flow, compared to treatment-as-usual with plaster cast, reduces VTE incidence and improves healing.

DETAILED DESCRIPTION:
The proposed intervention, intermittent pneumatic compression (IPC) is an evidence-based prevention for VTE in hospitalized patients and used in daily practice. IPC is, however, not currently used on outpatients and it is currently unknown if it reduces the risk of VTE during long term leg-immobilization. Plaster cast and orthosis treatments are currently used in daily practice on Achilles tendon ruptures and ankle fractures. At present there is no consensus about using VTE prophylaxis in leg-immobilized patients. Since pharmacoprophylaxis has shown low- or no VTE preventive effects in leg-immobilization, is not recommended by some guidelines.

Furthermore, since all patients will undergo clinical examinations and have DVT-screening performed with compression Doppler ultrasound (CDU) removal of leg immobilization this will comprise an extra security for the included patients to detect a VTE. If a VTE is detected clinical guidelines will be followed by initiating chemical VTE-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Acute unilateral Achilles tendon rupture or isolated Ankle Fracture
* Treatment starts within 10 days in a hospital setting

Exclusion Criteria:

* Inability or refusal to give informed consent for participation in the study
* Inability to comply with the study instructions
* Known kidney disorder
* Heart failure with pitting oedema
* Presence of known malignancy
* Current bleeding disorder
* Pregnancy
* Planned follow-up at another hospital
* Pilon fracture

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Venous Thromboembolic Events (VTE) | Up til the time of removal of leg immobilization, approx. 6-8 weeks
  The primary outcome is VTE defined as symptomatic Deep venous Thrombosis (DVT) or asymptomatic DVTs,or symptomatic pulmonary embolism

SECONDARY OUTCOMES:
Patient reported Outcome - ATRS | 6 months and 1 year
  symptoms will be assessed using the reliable and valid score; the Achilles tendon Total Rupture Score (ATRS)
Patient reported Outcome - FAOS | 6 months and 1 year
  symptoms will be assessed using the reliable and valid score; the Foot and Ankle Outcome Score (FAOS)
Patient reported Outcome - OMAS | 6 months and 1 year
  symptoms will be assessed using the reliable and valid score; the Olerud-Molander Ankle Score (OMAS)
Patient reported Outcome - EQ-5D-5L | 6 months and 1 year
  symptoms will be assessed using the reliable and valid score; EuroQol Group's questionnaire (EQ-5D-5L).
Functional outcome - muscular endurance tests (heel-rise) | 1 year
  Patient leg function will be measured by a validated endurance test (i.e. the heel-rise test) at 1 year post-injury.
Callus production | 6 weeks
  Microdialysis followed by quantification of procollagens will assess callus production in Achilles tendon healing.
VTE-preventive mechanisms | 6 weeks
  VTE-preventive mechanisms will be analyzed at the 6 week visit by assessments of profibrinolysis and coagulation factors as well as by blood-flow quantification .
Incidence of VTE in patients using low molecular weight heparin(LMWH) with or without adjvant IPC | 6-8 weeks
  Efficacy of LMWH with and without the use of IPC as to prevent VTE will be studied in order to confirm the efficency of a commonly used drug for VTE prophylaxis.
Patient mortality | 1year and 2 years
  Mortality of patients included will be recorded and investigated for cause of death. If the cause of death is VTE, this will be reported. The overall mortality rate in this study is expected to be low. Mortality will be investigated via patient journals at one year after study inclusion, and at 2 years via national mortality register.
Health economic analyses | 2 years
  Together with Karolinska Institutet, LIME, the trial treatment effects will involve a within-trial evaluation of cost effectiveness integrated into a decision-analytic model of longer run costs and health effects

CONTACTS AND LOCATIONS:
Overall Officials: Paul W Ackermann, MD, PhD, Principal Investigator — Karolinska University Hospital, 171 76 Stockholm, SWEDEN
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on reasonable requests.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After completion of the study.
Access Criteria: Data will be shared on reasonable requests to the steering committee.

REFERENCES:
- [Background] Arverud ED, Anundsson P, Hardell E, Barreng G, Edman G, Latifi A, Labruto F, Ackermann PW. Ageing, deep vein thrombosis and male gender predict poor outcome after acute Achilles tendon rupture. Bone Joint J. 2016 Dec;98-B(12):1635-1641. doi: 10.1302/0301-620X.98B12.BJJ-2016-0008.R1. PMID 27909125
- [Background] Domeij-Arverud E, Ackermann PW. Deep Venous Thrombosis and Tendon Healing. Adv Exp Med Biol. 2016;920:221-8. doi: 10.1007/978-3-319-33943-6_21. PMID 27535264
- [Background] Domeij-Arverud E, Labruto F, Latifi A, Nilsson G, Edman G, Ackermann PW. Intermittent pneumatic compression reduces the risk of deep vein thrombosis during post-operative lower limb immobilisation: a prospective randomised trial of acute ruptures of the Achilles tendon. Bone Joint J. 2015 May;97-B(5):675-80. doi: 10.1302/0301-620X.97B5.34581. PMID 25922463
- [Background] Abdul Alim M, Domeij-Arverud E, Nilsson G, Edman G, Ackermann PW. Achilles tendon rupture healing is enhanced by intermittent pneumatic compression upregulating collagen type I synthesis. Knee Surg Sports Traumatol Arthrosc. 2018 Jul;26(7):2021-2029. doi: 10.1007/s00167-017-4621-8. Epub 2017 Jul 1. PMID 28668970
- [Derived] Svedman S, Alkner B, Berg HE, Domeij-Arverud E, Jonsson K, Nilsson Helander K, Ackermann PW. STOP leg clots-Swedish multicentre trial of outpatient prevention of leg clots: study protocol for a randomised controlled trial on the efficacy of intermittent pneumatic compression on venous thromboembolism in lower leg immobilised patients. BMJ Open. 2021 May 20;11(5):e044103. doi: 10.1136/bmjopen-2020-044103. PMID 34016662
- See also: Official study site — http://ki.se/mmk/stop-leg-clots

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT03259204/Prot_SAP_000.pdf